CLINICAL TRIAL: NCT06276517
Title: Hidden Impairments During Subarachnoid Haemorrhage Recovery, Description and Evolution of a Newly Described Syndrom
Acronym: HIDDEN
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220918; 2022-A01739-34 (Other: IDRCB)
Record Dates: First submitted 2023-11-15; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Intracranial Hemorrhages
Keywords: post-HSA syndrome; subarachnoid hemorrhage
MeSH Terms: conditions — Intracranial Hemorrhages; Subarachnoid Hemorrhage | interventions — Surveys and Questionnaires; Coping Orientation to Problems Experienced Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with subarachnoid hemorrhage: Patients hospitalized in Lariboisière intensive care unit for subarachnoid hemorrhage
  Interventions: Other: questionnaire; Other: SS-QoL; Other: SF-36; Other: CIQ-R; Diagnostic Test: BREFF; Diagnostic Test: MoCA; Other: IADL; Other: mMRS; Other: PCL-5; Other: Brief-Cope

INTERVENTIONS:
Other: questionnaire — self-questionnaire with 16 questions, rated from 0 to 4, giving a total of 0 to 52 points.
  Other Names: Rivermead Post-Concussion symptoms questionnaire (RPQ)
Other: SS-QoL — 49-question self-administered questionnaire covering 12 domains (including work/productivity, mood, social roles, family roles, personality, etc.).
  Other Names: qustionnaire
Other: SF-36 — multidimensional, generic scale, i.e. one that assesses health status independently of causal pathology, sex, age and treatment
  Other Names: questionnaire
Other: CIQ-R — 16-question questionnaire with answers rated from 0 to 2 to assess Social reintegration
  Other Names: questionnaire
Diagnostic Test: BREFF — rapid frontal efficiency battery, 6 tests from 0 to 3 on each side
Diagnostic Test: MoCA — MoCA is a screening test for neurocognitive impairment. It comprises 11 categories scored from 0 to 6 for a total of 0 to 30 points.
Other: IADL — 8 questions rated from 0 to 1 to assess functional outcome
  Other Names: questionnaire
Other: mMRS — mMRS score from 0 to 4 to assess functional outcome
  Other Names: questionnaire
Other: PCL-5 — To assess the prevalence of post-traumatic stress using the PCL-5 self-questionnaire. PCL-5 is a 20-item self-administered questionnaire.
  Other Names: questionnaire
Other: Brief-Cope — 28-question self-questionnaires to study patients' coping strategies
  Other Names: questionnaire

SUMMARY:
Descriptive observational study in patients with spontaneous subarachnoid hemorrhage or following aneurysmal rupture to assess the presence of a post-HSA syndrome at 3 months, 6 months and 1 year, and its impact on functional outcome using the Rivermead questionnaire

DETAILED DESCRIPTION:
Every year, subarachnoid hemorrhage affects 9.1 people per 100,000 worldwide, with a peak between the ages of 50 and 60. Its frequency and relatively young age of onset make it a major source of decline in healthy life years.

Progress over the past thirty years has led to a 57% reduction in mortality, but these figures do not always reflect the day-to-day reality of these patients, for whom recovery remains incomplete in almost half of cases. For example, a third of patients have not returned to work at one year, and of those who have, only half have returned to work full-time. In 2020, a Norwegian team showed that, at one year, a third of patients suffer from a "post-HSA syndrome", as yet little described, but which seems very similar to the post-concussion syndrome experienced by patients after head trauma. In their study, only 3% of patients with this syndrome returned to work at one year. A better understanding of the incidence of this syndrome, as well as its evolution and determinants, is therefore essential.

With this in mind, the investigators chose to assess the presence of post-SAH syndrome at 3 months and its repercussions on return to work, using the Rivermead questionnaire.

Secondly, in view of the prevalence of post-traumatic stress syndrome at 3 years (a quarter of patients), the investigators wished to study the factors determining the presence of post-HSA syndrome and an inability to return to work at 3 months, 6 months, 1 year.

ELIGIBILITY:
Inclusion Criteria:

Patient aged 18 to 65

* Patient hospitalized in intensive care unit at Hôpital Lariboisière between September 2022 and September 2023 for subarachnoid hemorrhage due to aneurysmal rupture.
* Patient affiliated to the French social security system
* Patient expressing no objection

Exclusion Criteria:

* Motor deficits persisting 1 month after SAH
* Hospitalization > 1 month
* Patient does not speak French
* Patient with diagnosis of neurodegenerative disease.
* Traumatic meningeal hemorrhage
* Patients on AME

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 65 who had presented with an episode of spontaneous subarachnoid haemorrhage or aneurysmal rupture, excluding meningeal haemorrhage due to trauma,
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the presence of post SAH syndrome at 3 months and its impact on return to work using the Rivermead Post-Concussion symptoms questionnaire (RPQ), and its impact on functional outcome. | 3 months
  The Rivermead questionnaire is a 16-item self-administered questionnaire, rated from 0 to 4, giving a total of 0 to 52 points.
  This scale was created to assess post-concussion syndrome, which in many ways is similar to what patients experience after a SAH.
  The higher the score, the greater the difficulties experienced by the patient. A score of 3 or 4 for any of the responses indicates that the patient is incapacitated.

SECONDARY OUTCOMES:
- study the factors determining the presence of a post-HSA syndrome and an inability to return to work at 3 months, 6 months and 1 year | 3 months, 6 months and 1 year,
  Quality of life assessed using the SS-QoL questionnaire, specific to stroke patients. Self-questionnaire with 49 questions covering 12 domains (including work/productivity, mood, social roles, family roles, personality).
To study the prevalence of post-traumatic stress in this population | 3 months, 6 months and 1 year,
  Assess the prevalence of post-traumatic stress in this population using the PCL-5 self-questionnaire. PCL-5 is a 20-question self-questionnaire.
Study patients' coping strategies in relation to functional recovery using the Brief-Cope self-questionnaire | 3 months, 6 months and 1 year,
  Brief-Cope self-questionnaire (28-question self-questionnaires).

IPD SHARING:
Plan to Share IPD: No